CLINICAL TRIAL: NCT03199131
Title: The Right Ventricle in Chronic Pressure Overload: Identifying Novel Molecular Targets for Functional Imaging
Acronym: MVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-A00149-40
Record Dates: First submitted 2017-03-22; First posted 2017-06-26 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTEPH (Experimental): Patients undergoing pulmonary endarterectomy for the treatment of chronic thromboembolic pulmonary hypertension (CTEPH).
  Interventions: Procedure: Right ventricular biopsies
- Control group (Other): Patients undergoing adult cardiac surgery without evidence of pulmonary hypertension.
  Interventions: Procedure: Right ventricular biopsies

INTERVENTIONS:
Procedure: Right ventricular biopsies — a right ventricular biopsy will be taken intraoperatively during either pulmonary endarterectomy (experimental group) or open cardiac surgery (control group).

SUMMARY:
Chronically elevated pulmonary pressures do not immediately result in right ventricular failure. During the initial period of exposure, the RV adapts to the increased afterload by altering its metabolism and morphology so as to meet the increased work requirement. Several, interconnected adaptive mechanisms have been proposed, including myocyte hypertrophy, a switch in the primary fuel used for ATP generation, increased angiogenesis, and decreased production of mitochondrial reactive oxygen species. While adaptation is initially successful in many cases, it is temporary, and after an uncertain period of time, the ventricle begins to fail. This transition from a compensated to decompensated state is difficult to predict clinically, and patients with different etiologies of CPOS progress to overt RV failure over significantly different time periods. This variability hinders the implementation of treatments that are tailored to a specific disease stage.

DETAILED DESCRIPTION:
Chronically elevated pulmonary pressures do not immediately result in right ventricular failure. During the initial period of exposure, the RV adapts to the increased afterload by altering its metabolism and morphology so as to meet the increased work requirement. Several, interconnected adaptive mechanisms have been proposed, including myocyte hypertrophy, a switch in the primary fuel used for ATP generation, increased angiogenesis, and decreased production of mitochondrial reactive oxygen species. While adaptation is initially successful in many cases, it is temporary, and after an uncertain period of time, the ventricle begins to fail. This transition from a compensated to decompensated state is difficult to predict clinically, and patients with different etiologies of CPOS progress to overt RV failure over significantly different time periods. This variability hinders the implementation of treatments that are tailored to a specific disease stage. As right heart failure is the primary outcome determinant in patients with pulmonary hypertension, understanding the major mediators of RV compensation, failure and recovery is essential to improving patient survival. Recently, there have been significant advances in the ability to assess RV function in vivo using functional imaging techniques, including positron emission tomography (PET) and cardiac MRI (CMR). CMR is an established and validated method of precisely defining cardiac structure and function, and new PET protocols have been developed that measure glucose utilization, oxygen consumption, apoptosis and angiogenesis. Importantly, the in vivo nature of PET and CMR allow for the non-invasive collection of detailed structural, metabolic and physiologic data on the performance of the RV5. When taken in combination with established echocardiographic evaluation, these new platforms allow in-depth analysis of cardiac structure and function without the need for invasive procedures. In order to maximize the potential of these techniques, however, a molecular imaging target needs to be identified so as to allow physicians to detect the transition from a compensated to decompensated state. Such a marker has not yet been reported

ELIGIBILITY:
-Inclusion Criteria:

Chronic thromboembolic pulmonary hypertension group:

* Patients undergoing pulmonary endarterectomy at Marie Lannelongue Surgical Center for the treatment of chronic thromboembolic pulmonary hypertension.

Control group:

* Patients undergoing adult cardiac surgery without evidence of pulmonary hypertension on preoperative assessment
* Exclusion Criteria:

Chronic thromboembolic pulmonary hypertension group:

* Insufficient biopsy material,
* pre-operative therapy with bosentan or sildenafil

Control group:

* Insufficient biopsy sample,
* ischemic cardiomyopathy,
* miral or tricuspid valve disease,
* pre-operative pulmonary hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
relationship between the metabolic, morphologic and functional alterations in the right ventricle | to investigate the relationship between the metabolic, morphologic and functional alterations in the right ventricle before surgery,one and six months after surgery.

SECONDARY OUTCOMES:
validation in human subjects of metabolic signaling pathway alterations found in animal model | analyse gene and protein expression during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Mercier, MD, PhD, Principal Investigator — Marie Lannelongue Hospital
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No